CLINICAL TRIAL: NCT01982513
Title: Influence of the Method of Alleviation of Aorto-Caval Compression on the Trans-Hepatic Ultrasound-Assessed Inferior Vena Cava Diameter In Pregnant Patients: An Observational Study of the Left Lateral Tilt and of the Left Uterine Displacement
Brief Title: Influence of the Method of Alleviation of Aorto-Caval Compression on the Trans-Hepatic Ultrasound-Assessed Inferior Vena Cava Diameter In Pregnant Patients
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13-09
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Pregnancy; Cardiac Arrest
Keywords: Cardiopulmonary Resuscitation; Pregnancy; Ultrasound; Inferior Vena Cava
MeSH Terms: conditions — Heart Arrest | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Term pregnant patients: ASA I-II term (36-40 weeks) non-laboring women with singleton pregnancies who are admitted at MSH for induction of labor, elective cesarean section or for observation for any medical reason.
  These patients will be examined in 4 positions with the ultrasound.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — The IVC will be visualized and images obtained using the intercostal window in both longitudinal and transverse planes.

SUMMARY:
Cardiac arrest during pregnancy is rare but may result in poor maternal and fetal outcome. Because of its rare occurrence and ethical issues this topic is not very well studied and many questions pertaining to maternal resuscitation remain unanswered. One of the challenging aspects of cardiopulmonary resuscitation in a term pregnant patient is the ideal positioning during chest compressions. International societies have made recommendations regarding management of pregnant patients during cardiac arrest. They advocate the use of left lateral position with 30 degrees tilt or manual uterine displacement. However these recommendations are not based on high level of evidence. Ultrasound has been used to visualize the change in diameter of great vessels to determine the volume status or adequacy of blood circulation of these patients. This approach can be used to study the adequacy of blood circulation of pregnant patients in different positions. The objective of this study is to compare the change in Inferior vena cava diameter obtained with pregnant women in either the left lateral tilt or in the supine position with a manual uterine displacement, compared to the left lateral position and the supine position.

Our hypothesis is that the inferior vena cava diameter obtained in the supine position with manual left uterine displacement would be larger as compared to that obtained with women positioned with a 30-degree tilt.

DETAILED DESCRIPTION:
Using the non-invasive technology of ultrasound we will be able to determine the degree of aorto-caval compression in pregnant women placed in different positions. The results of this study will help us to determine the optimal patient positioning for each individual. This in future may help us in improving outcomes not only during labor and anesthesia, but also during maternal resuscitation in critical cases.

The results of this study will help us to determine the best technique to minimize aorto-caval compression in the term pregnant patient. The results of this study will be useful to establish firm maternal resuscitation guidelines. We will be able to determine the optimal maternal position during cardiopulmonary resuscitation and this may improve both maternal and fetal resuscitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Term pregnancy (36-40 weeks)
* Singleton pregnancy

Exclusion Criteria:

* Patients with known cardiac disease, severe preeclampsia on medication
* Multiple gestation
* Breech presentation
* Patients unable to comply with the 4 positions (left lateral, left tilt, supine and supine with manual displacement)
* Patients unable or unwilling to consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non-laboring, term prengnant women with singleton pregnancies who are admitted at Mount Sinai Hospital for induction of labor, elective cesarean section or for observation for any medical reason.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
IVC maximum diameter | 20 minutes
  The IVC maximum diameter in each position (measured during expiration).

SECONDARY OUTCOMES:
Fetal Heart Rate | 20 minutes
  The fetal heart rate will be monitored during the last minute of observation in each position.
Maternal vitals | 20 minutes
  Maternal blood pressure and heart rate will be monitored during the last minute of observation in each position.
IVC minimum diameter | 20 minutes
  The IVC minimum diameter in each position (measured during inspiration).
IVC Index | 20 minutes
  IVC index (IVI) = IVC(max)-IVC (min)/IVC(max)

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada